CLINICAL TRIAL: NCT02332213
Title: Volatile Marker Testing for Digestive Cancer and Precancerous Lesion Detection, Evaluation of Confounding Factors
Brief Title: Volatile Markers in Digestive Cancer
Acronym: VOLGACORE
Status: Completed | Type: Observational
Sponsor: University of Latvia (Other)
Collaborators: Technion, Israel Institute of Technology (Other); Lithuanian University of Health Sciences (Other); Karolinska Institutet (Other); German Cancer Research Center (Other); Digestive Diseases Centre GASTRO (Other); Riga East Clinical University Hospital (Other Government); Academic Histology Laboratory (Latvia) (Other); JLM Innovation GmbH (Germany) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2914; LZP Nr. 2014.10-5 (Other: Latvian Research Council)
Record Dates: First submitted 2014-12-30; First posted 2015-01-06 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer; Colorectal Adenoma; Gastric Cancer; Peptic Ulcer Disease; Atrophic Gastritis; Intestinal Metaplasia; H.Pylori Infection; Normal Control; Average-risk General Population
Keywords: Volatile organic compounds; Nanosensor technology; GC-MS; Breath-testing; Digestive cancer; Precancerous lesions; Colorectal cancer; Adenoma; Gastric cancer; Atrophic gastritis; OLGIM
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Peptic Ulcer; Gastritis, Atrophic; Gastrointestinal Neoplasms; Adenoma | interventions — Gastroscopy; Biopsy; Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Exhaled air samples being stored in specific adsorbent media Plasma/serum samples for group stratification Faecal samples for occult blood testing and microbiota analysis Biopsy samples from stomach and colon
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (9):
- 1. Colorectal cancer: Patients with histologically confirmed colorectal cancer (adenocarcinoma)
  Interventions: Procedure: Breath sampling for volatile marker detection; Procedure: Colonoscopy with biopsies or lesion removal when required; Procedure: Plasma/serum sampling; Procedure: Faecal sample acquisition; Procedure: Histological evaluation of the surgery material
- 2. Colorectal high-risk lesions: Patients without colorectal adenocarcinoma, but carrying high-risk adenomatous polyps being described by one of the following: 1) size≥1 cm; 2) high-grade dysplasia; 3) villous component. Prior to removal of the lesions.
  Interventions: Procedure: Breath sampling for volatile marker detection; Procedure: Colonoscopy with biopsies or lesion removal when required; Procedure: Plasma/serum sampling; Procedure: Faecal sample acquisition
- 3. Colorectal low-risk adenoma: Patients without colorectal adenocarcinoma and without colorectal high-risk lesions as described under Group 2 criteria
  Interventions: Procedure: Breath sampling for volatile marker detection; Procedure: Colonoscopy with biopsies or lesion removal when required; Procedure: Plasma/serum sampling; Procedure: Faecal sample acquisition
- 4. Group of control (colorectal): Patients having undergone colonoscopy without an evidence for colorectal lesions fulfilling Group 1 or Group 2 or Group 3 criteria. Prior to removal of the lesions.
  Interventions: Procedure: Breath sampling for volatile marker detection; Procedure: Colonoscopy with biopsies or lesion removal when required; Procedure: Plasma/serum sampling; Procedure: Faecal sample acquisition
- 5. Gastric cancer: Patients with histologically confirmed gastric cancer (adenocarcinoma)
  Interventions: Procedure: Breath sampling for volatile marker detection; Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Faecal sample acquisition; Procedure: Histological evaluation of the surgery material
- 6. Gastric dysplasia: Patients without gastric adenocarcinoma but with histologically confirmed dysplasia (either high- or low-grade) of the stomach
  Interventions: Procedure: Breath sampling for volatile marker detection; Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Faecal sample acquisition
- 7. High-risk gastric lesions: Patients graded Stage III-IV according to OLGIM (Operative Link of Gastric Intestinal Metaplasia Assessment) staging system, but excluding those with dysplasia (Group 5)
  Interventions: Procedure: Breath sampling for volatile marker detection; Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Faecal sample acquisition
- 8. Normal and low-risk gastric lesions: Staged 0-III according to OLGIM. Dysplasia should be excluded
  Interventions: Procedure: Breath sampling for volatile marker detection; Procedure: Upper endoscopy with biopsies; Procedure: Plasma/serum sampling; Procedure: Faecal sample acquisition
- 9. Average risk population: Average risk population of both genders aged 40-64 at the time of inclusion lacking alarm symptoms for gastrointestinal cancer.
  Interventions: Procedure: Breath sampling for volatile marker detection; Procedure: Plasma/serum sampling; Procedure: Faecal sample acquisition

INTERVENTIONS:
Procedure: Breath sampling for volatile marker detection — Acquisition of two exhaled breath samples of alveolar air to be analysed by GCMS and nanosensor technology
Procedure: Upper endoscopy with biopsies — Upper endoscopy with proper biopsy work-up will be used for identification and stratification of gastric lesions as well as acquisition of biopsies for microbiota testing
  Groups: 5. Gastric cancer; 6. Gastric dysplasia; 7. High-risk gastric lesions; 8. Normal and low-risk gastric lesions
Procedure: Colonoscopy with biopsies or lesion removal when required — Colonoscopy with proper biopsy or polypectomy material work-up will be used for identification and stratification of colorectal lesions as well as acquisition of biopsies for microbiota testing
  Groups: 1. Colorectal cancer; 2. Colorectal high-risk lesions; 3. Colorectal low-risk adenoma; 4. Group of control (colorectal)
Procedure: Plasma/serum sampling — Plasma/serum sampling will be used to obtain information for group stratification, e.g. H.pylori status determination
Procedure: Faecal sample acquisition — Faecal samples will be obtained for faecal occult blood testing as well as microbiota analysis
Procedure: Histological evaluation of the surgery material — The material obtained during surgery (stomach or colorectal) will be used for confirmation of the diagnosis in cancer groups. Surgery itself will be performed according to the clinical indications, and will not be extended (i.e. cannot be considered a study intervention)
  Groups: 1. Colorectal cancer; 5. Gastric cancer

SUMMARY:
The study is aimed to determine the potential of volatile marker testing for identification of gastrointestinal cancers (in particular - colorectal and gastric cancers), the related precancerous lesions in the stomach and colon.

The study will be addressing the role of confounding factors, including lifestyle factors, diet, smoking as well as addressing the potential role of microbiota in the composition of exhaled volatile markers.

DETAILED DESCRIPTION:
Patients with established disease (cancer, precancerous lesions) as well as patients investigated for the lesions and having been documented lack of the lesions will be enrolled to the study at clinical sites in Europe (Latvia, Lithuania). In addition, group of persons from general population at average risk for developing the target disease will be also enrolled.

Testing of volatile markers will be conducted by one of two methods: 1) gas chromatography coupled to mass spectroscopy (GS-MS) and 2) nanosensor technology.

Volunteers (including patients with established disease) will be enrolled prior the removal of the target lesion (e.g. surgery for cancer or polypectomy in the case of a polyp).

The study will be conducted by utilizing the experience of institutions in the European Union and Israel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with verifies colorectal cancer (Group 1)
* Patients with verified gastric cancer (Group 5)
* Patients undergoing colonoscopy due to clinical indications (group 2-4)
* Patients undergoing upper endoscopy due to clinical indications (Group 6-8)
* Average-risk population group aged 40-64 at inclusion without alarm symptoms (Group 9)
* Motivation to participate in the study
* Physical status allowing volatile marker sampling and other procedures within the protocol
* Signed consent

Exclusion Criteria:

* Known other active cancer
* Ventilation problems, airway obstruction
* Unwillingness or inability to co-operate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer patients (Group 1 and 5) will be predominantly enrolled at the time scheduled for surgery, however also patients undergoing diagnostic procedures (endoscopy) will be eligible
  Patients without malignant disease but defined colorectal (Groups 2-4) status will be predominantly enrolled prior colonoscopy in out-patient settings. Sampling starting from 1 week after colonoscopy will be allowed if the lesions will not get removed during the index endoscopy
  Patients without malignant disease but defined gastric mucosal status (Groups 6-8) status will be predominantly enrolled prior upper endoscopy in out-patient settings. Sampling starting from 2 days after upper endoscopy will be allowed if the lesions will not get removed during the index endoscopy
  Average cancer risk subjects (Group 9) will get enrolled by inviting individuals predominantly selected from the lists of general practitioners.
Sampling Method: Non-Probability Sample
Enrollment: 2022 (Actual)
Dates: Start 2014-01; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Performance of nanoarray sensor testing to detect target lesions | At the time of breath sampling
  Sensitivity, specificity, overall accuracy of nanoarray sensor testing for VOCs to detect the target lesions in the blinded analysis
VOCs differentiating the study groups | At the time of breath sampling
  List of VOCs assayed by GC-MS with statistical difference between the study groups

SECONDARY OUTCOMES:
Identification of characteristic VOC pattern in risk age groups | At the time of sampling
  List of characteristic VOCs in general population at risk for developing gastrointestinal cancer, including analysis of confounding factors, e.g. dietary habits, smoking, and profession.
VOC pattern changes following treatment | At baseline and every 6 months within 3 year period
  Significant change in VOC content before and following treatment (surgery, medical therapy, combined)
Groups of gastrointestinal microbiota correlating to VOCs | At the time of sampling
  List of gastrointestinal microbiota groups (phylum/genus level) with positive correlation to particular VOCs

OTHER OUTCOMES:
VOC pattern changes following intervention to microbiota | At baseline and following the intervention (1 week, 1 month)
  Significant change in VOC content before and following intervention upon microbiome (antibiotic intake, colon cleansing)
Gastric microbiome changes following intervention to microbiota | At baseline and 3 years after intervention
  Significant change in gastric microbiome (phyla, genera) before and following intervention upon microbiome (antibiotic intake)
Gastrointestinal microbiome in cancer patients | At the time of sampling
  Significant differences in the composition of gastric and colonic microbiome (phyla, genera) in cancer patients, patients with precancerous lesions and controls

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Haick, Ph.D., Principal Investigator — Technion, Israel Institute for Technology (Israel)
Locations (2):
- University of Latvia, Riga, Latvia
- Lithuanian University of Health Sciences, Kaunas, Lithuania

REFERENCES:
- [Background] Haick H, Broza YY, Mochalski P, Ruzsanyi V, Amann A. Assessment, origin, and implementation of breath volatile cancer markers. Chem Soc Rev. 2014 Mar 7;43(5):1423-49. doi: 10.1039/c3cs60329f. Epub 2013 Dec 4. PMID 24305596
- [Background] Xu ZQ, Broza YY, Ionsecu R, Tisch U, Ding L, Liu H, Song Q, Pan YY, Xiong FX, Gu KS, Sun GP, Chen ZD, Leja M, Haick H. A nanomaterial-based breath test for distinguishing gastric cancer from benign gastric conditions. Br J Cancer. 2013 Mar 5;108(4):941-50. doi: 10.1038/bjc.2013.44. PMID 23462808
- [Background] Amal H, Leja M, Broza YY, Tisch U, Funka K, Liepniece-Karele I, Skapars R, Xu ZQ, Liu H, Haick H. Geographical variation in the exhaled volatile organic compounds. J Breath Res. 2013 Dec;7(4):047102. doi: 10.1088/1752-7155/7/4/047102. Epub 2013 Nov 1. PMID 24184568